CLINICAL TRIAL: NCT06716294
Title: Effectiveness Of Radiofrequency Ablation And Stabilization In Metastatic Spine Lesions By PET Confirmation
Acronym: ABLASPINE
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexis Kelekis, PROFESSOR OF DIAGNOSTIC AND INTERVENTIONAL RADIOLOGY, National and Kapodistrian University of Athens
Other Study IDs: 46351/2020
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Bone Cancer Metastatic; Radiofrequency Ablation; Spine Metastases; Vertebral Metastasis
MeSH Terms: interventions — Radiofrequency Ablation; Vertebroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Radiofrequency Ablation and Bone Augmentation — Percutaneous Tumor Ablation of Spine Lesions followed by Polymer Augmentation
  Other Names: Vertebroplasty

SUMMARY:
This pilot study will try to demonstrate metabolic changes in spine lesions treated by Augmentation and Ablation, according to existing standards of practice. Our purpose is to show the efficacy of a new radiofrequency radioablation (RFA) in combination with augmentation, using a percutaneous ablation device (Osteocool-Medtronic) in the treatment of secondary vertebral bone tumor, avoiding concurrent bias related to other treatments of the disease.

DETAILED DESCRIPTION:
Only patient supposed to undergo percutaneous vertebral augmentation for secondary osteolytic and mixed (lytic and sclerotic) spine tumors with one to three active lesions will be enrolled. Lesions to be treated must be metabolically active on PET-CT, performed during the last month. Patients will be informed and sign and inform consent. Patients will be treated with Augmentation and Ablation (Osteocool-Medtronic). Post treatment patients will be submitted to a new PET-CT in order to verify activity on treated site.

ELIGIBILITY:
Inclusion Criteria:

* only patients with secondary osteolytic and mixed (lytic and sclerotic) spine tumors with one to three active lesions will be enrolled.
* lesions to be treated must be metabolically active on PET-CT performed during the last month.
* Patients will be informed and sould sign an inform consent.
* post treatment patients should submittes a new PET-CT in order to verify the activity of the treated area.

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Sixteen (16) patients will be enorolled.
  * - only patients with secondary osteolytic and mixed (lytic and sclerotic) spine tumors with one to three active lesions will be enrolled.
  * lesions to be treated must be metabolically active on PET-CT performed during the last month.
  * Patients will be informed and sould sign an inform consent.
  * post treatment patients should submittes a new PET-CT in order to verify the activity of the treated area.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PET | SUV measurement of PET in 24 hours
  PET ACTIVITY

SECONDARY OUTCOMES:
GBPI | 1 MONTH, 6 MONTHS, 12 MONTHS
  NVS SCORE OF PAIN AND MOBLITY

CONTACTS AND LOCATIONS:
Overall Officials: ALEXIOS KELEKIS, MD, PHD, Principal Investigator — National and Kapodistrian University of Athens, Greece
Locations (1):
- Attikon General University Hospital, Athens, Haidari, Greece

IPD SHARING:
Plan to Share IPD: Undecided